CLINICAL TRIAL: NCT02534090
Title: Evaluation of Feeding Intolerance in Premature Infants Using Near Infrared Spectroscopy
Acronym: NIRS/NICU2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ricardo Castillo-Galvan, MD, Newborn Medicine Department, Brigham and Women's Hospital
Other Study IDs: 2015P001806
Record Dates: First submitted 2015-08-23; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Feeding Intolerance; Necrotizing Enterocolitis; Premature Infant
Keywords: Premature; Preterm; Necrotizing; Enterocolitis; NIRS
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth; Enterocolitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Feeding Intolerant Preterm Infants: 32 weeks to 36 weeks 6 days old of post menstrual age infants, feeding intolerants monitored with INVOS device for rSO2
- Feeding Tolerant Preterm Infants (Controls): 32 weeks to 36 weeks 6 days old of post menstrual age infants without problems through the enteral feedings.

SUMMARY:
Nowadays feeding intolerance (FI) is a common condition among preterm infants. It has been estimated that 16%-29% of premature infants admitted to neonatal intensive care units (NICUs) develop feeding intolerance at some point during their length of stay. The most frequent signs of FI are the presence of abdominal distension, abundant and/or bilious gastric residuals and vomiting suggesting an inability of the infant to further tolerate enteral nutrition, it increases with decreasing in gestational age (GA) and birth weight (BW). FI represents one of the most uncontrollable variables in the early nutritional management of these infants, and may lead to suboptimal nutrition, delayed attainment of full enteral feeding and prolonged parenteral nutrition supply.

NIRS has been used in preterm infants to evaluate changes in cerebral perfusion and oxygenation. It provides real time insight into the oxygen delivery, presented as regional oxygen saturation rSO2 with lower values than SpO2 distal pulse-oximetry where is mostly measured as arterialized capillary bed (around 55% vs 98% Oxygen saturation in regional NIRS vs conventional pulse-oximetry). Light easily penetrates the thin tissues of the neonate through bone and soft tissue, particularly the thin capillary bed of the tissues; NIRS provides non-invasive, continuous information on tissue perfusion and oxygen dynamics.

This technique uses principles of optical spectrophotometry that make use of the fact that biological material, including the skull, is relatively transparent in the NIR range.

Dave et al. evaluated the abdominal tissue oxygenation with NIRS, and showed that preterm infants change their cerebral - splanchnic oxygenation ratios during feedings, mainly because an increasing in the splanchnic oxygenation.

Gay et al. performed abdominal NIRS in premature piglets showing association of perfusion/oxygen changes with NEC spectrum.

The investigators would like to evaluate the association between feeding intolerance and unchanged splanchnic regional saturation and variation in the cerebral splanchnic ratio.

Innovation:

FI diagnosis follows a subjective approach, where the clinician is worried in further risk of develop Necrotizing enterocolitis (NEC). This non-studied relationship (FI and NEC) lower the threshold for the diagnosis of FI. Furthermore, infants with FI diagnosis commonly are subject of stop or slow the progression of feedings, increasing the risk of intestinal villi atrophy, and increase the length of parenteral nutrition support, and also the length of stay in the NICU settings. If NIRS technology help the clinicians to detect true abnormalities objectively as a new monitor assessing adequate feeds progress decreasing failure to feed, and therefore diminishing the need for parenteral feeds and further complication associated with it.

DETAILED DESCRIPTION:
Approach Basic study design The study design is a matched-pair case-control cohort, longitudinal.

Study population and assembly of patients Premature infants from 32 to 36 6/7 weeks of postmenstrual age, with feeding tolerance at least of 50ml/kg/day, inpatients at the Brigham and Women's NICU.

Inclusion criteria:

* Premature infants from 32 to 36 6/7 weeks of postmenstrual age, with feeding tolerance at least of 50ml/kg/day which have been diagnosed with food intolerance.
* Control group will be composed with patients from the same population age range tolerating at least 50 ml/Kg/day (Half of the minimum full feeds daily requirement) of Human milk of enteral Formula delivered in bolus, 6 to 8 times per day.
* Written informed consent from parent(s) or guardian.

Exclusion criteria:

* Premature infants with know conditions that could affect the attachment of the sensors in the body areas as Gastroschisis, Omphalocele, Post surgical intestine resection, on peritoneal dialysis, with lacerations in the abdomen and frontal area of the head.
* Infants who have been diagnosed with Necrotizing enterocolitis.
* Infants with current diagnosis of Sepsis and/or Systemic Inflammatory Response Syndrome (SIRS).
* Infants with severe Intra-Ventricular Hemorrhage (Intra-cranial Hemorrhage).
* Infants with Hereditary Spherocytosis, total or partial (hypoplasia) congenital asplenia hypoplasia.

Exposures and their measurement The investigators will use two NIRS devices, the INVOS™ 5100c Cerebral/Somatic Oximeter is a 2 wavelength, diffuse reflectance spectroscopy system employing near infrared light to estimate the percentage of hemoglobin saturated with oxygen in tissue underneath the sensor. An adhesive sensor containing a light source and 2 photodiodes is applied to the skin over the tissue of interest and the returning light is analyzed for oxyhemoglobin and deoxyhemoglobin light absorption. Absorption signals from the photodiode closer to the light source are subtracted from those from the farther photodiode where the returning photons penetrate more deeply in the tissue. This suppresses absorption events originating in the outer layers of tissue that are common to both photodiodes, including the effects of skin pigmentation and subcutaneous tissues. This method of "spatial resolution" also allows estimation of scattering to improve measurement accuracy.

This is a non-invasive device Food and Drug Administration (FDA) approved (FDA 510k #K082327), with an intended use for infants with a weight greater than 2.5 Kg. Given that the target population of this study has weights under the description to use, and being used in cerebral oxygen monitoring, in order to be approved by the Institutional Board Review (IRB) committee. The investigators will catalogue it as non-significant risk device under the Investigational Device Exemption (IDE), 21 CFR 812.

The device has four channels where the light sensors will retrieve the lectures from the splanchnic (left flank), mesenteric (infra-umbilical), muscular (either right or left thigh) and cerebral (forehead) areas. The NIRS sensors Cerebral (IS-C) and Somatic (IS-S) Infant/Neonatal Somatic OxyAlert® will be attached directly to the infant skin in order to obtain the area lecture.

The cases will be diagnosed as feeding intolerant for the attending physician staff and those patients that have been at least with 50ml/Kg/day in their enteral feedings will be approached.

Once the case is attached with the NIRS device, the selection of the matching control will take place, a feeds tolerating infant (at least 50 mL/Kg/day) sharing gestational range age and gender if possible. for The study coordinators will obtain the consent from the parent(s); those families will have the opportunity to speak with the Physician investigator (PI). All the staff members are certified in the CITI program (Collaborative IRB Training Initiative) to ensure and discuss the protocol with the infant's parent(s) or guardian. After the sensors have been attached the data will be recorded the display of the monitor will be turned off, the data will be extracted and analyzed.

Confounders and their measurement The study design will allow to minimize the confounders with restriction (inclusion and exclusion criteria), same at risk population, and matching the cases.

Low perfusion status need to be assessed monitoring vital signs (HR,RR,BP) and pulse-oximetry (SpO2).

Outcomes and their measurement Clinical outcome data will be correlated with tissue oxygen saturation (TOI) from the NIRS device, other outcomes variables include: length of NICU stay, morbidity, mortality, feeding tolerance, advance in the feedings and abdominal sign of intolerance, abdominal distension, gastric residues greater than 50% of the intermittent bolus. Other variables will be recorded, infant perinatal history, level of oxygen requirements, ventilatory support status, morbidities associated, laboratory studies, vital signs and parenteral nutrition status. oxygen saturation by standard pulse oximetry, formula and/or human milk feeding status, and follow them until their discharge from the Hospital, looking for length of stay, development of Necrotizing enterocolitis, and/or Broncho-pulmonary dysplasia. The data will be extracted from their clinical records (EPIC System).

ELIGIBILITY:
Inclusion Criteria:

* Premature infants from 32 to 36 6/7 weeks of postmenstrual age, with feeding tolerance at least of 50ml/kg/day which have been diagnosed with food intolerance.
* Control group will be composed with patients from the same population age range tolerating at least 50 ml/Kg/day (Half of the minimum full feeds daily requirement) of Human milk of enteral Formula delivered in bolus, 6 to 8 times per day.
* Written informed consent from parent(s) or guardian.

Exclusion Criteria:

* Premature infants with know conditions that could affect the attachment of the sensors in the body areas as Gastroschisis, Omphalocele, Post surgical intestine resection, on peritoneal dialysis, with lacerations in the abdomen and frontal area of the head.
* Infants who have been diagnosed with Necrotizing enterocolitis.
* Infants with current diagnosis of Sepsis and/or Systemic Inflammatory Response Syndrome (SIRS).
* Infants with severe Intra-Ventricular Hemorrhage (Intra-cranial Hemorrhage). Infants with Hereditary Spherocytosis, total or partial (hypoplasia) congenital asplenia hypoplasia.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature infants from 32 weeks to 36 weeks 6 days of post menstrual age.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Low abdominal (Splanchnic) tissue oxygenation (less than 0.50 Oxygen saturation). | 3 days
  There is not an specific threshold of regional oxygen saturation measured through NIRS, the investigators want to evaluate the range of saturation as follows: 1. Greater than 0.60; 2. .50 to .60 and less than 0.50 Oxygen saturation, reading above expected, expected, below expected respectively.

SECONDARY OUTCOMES:
Cerebral Splanchnic Ratio (CSOR) < 0.75 | 3 days
  NIRS Cerebral Oxygenation and Splanchnic Oxygenation help to obtain an index where 0.75 to 0.95 could be considering adequate and below 0.75 considered abnormal. Area under the ROC curve is needed.

REFERENCES:
- [Background] Murkin JM, Arango M. Near-infrared spectroscopy as an index of brain and tissue oxygenation. Br J Anaesth. 2009 Dec;103 Suppl 1:i3-13. doi: 10.1093/bja/aep299. PMID 20007987
- [Result] Dani C, Corsini I, Generoso M, Gozzini E, Bianconi T, Pratesi S. Splanchnic Tissue Oxygenation for Predicting Feeding Tolerance in Preterm Infants. JPEN J Parenter Enteral Nutr. 2015 Nov;39(8):935-40. doi: 10.1177/0148607114538671. Epub 2014 Jun 16. PMID 24934405
- [Result] Fanaro S. Feeding intolerance in the preterm infant. Early Hum Dev. 2013 Oct;89 Suppl 2:S13-20. doi: 10.1016/j.earlhumdev.2013.07.013. Epub 2013 Aug 17. PMID 23962482
- [Result] Wolfberg AJ, du Plessis AJ. Near-infrared spectroscopy in the fetus and neonate. Clin Perinatol. 2006 Sep;33(3):707-28, viii. doi: 10.1016/j.clp.2006.06.010. PMID 16950321
- [Result] Pellicer A, Bravo Mdel C. Near-infrared spectroscopy: a methodology-focused review. Semin Fetal Neonatal Med. 2011 Feb;16(1):42-9. doi: 10.1016/j.siny.2010.05.003. Epub 2010 Jun 26. PMID 20580625
- [Result] Wolf M, Greisen G. Advances in near-infrared spectroscopy to study the brain of the preterm and term neonate. Clin Perinatol. 2009 Dec;36(4):807-34, vi. doi: 10.1016/j.clp.2009.07.007. PMID 19944837
- [Result] Patel J, Marks K, Roberts I, Azzopardi D, Edwards AD. Measurement of cerebral blood flow in newborn infants using near infrared spectroscopy with indocyanine green. Pediatr Res. 1998 Jan;43(1):34-9. doi: 10.1203/00006450-199801000-00006. PMID 9432110
- [Result] Yoxall CW, Weindling AM, Dawani NH, Peart I. Measurement of cerebral venous oxyhemoglobin saturation in children by near-infrared spectroscopy and partial jugular venous occlusion. Pediatr Res. 1995 Sep;38(3):319-23. doi: 10.1203/00006450-199509000-00008. PMID 7494653
- [Result] Pellicer A, Gaya F, Madero R, Quero J, Cabanas F. Noninvasive continuous monitoring of the effects of head position on brain hemodynamics in ventilated infants. Pediatrics. 2002 Mar;109(3):434-40. doi: 10.1542/peds.109.3.434. PMID 11875138
- [Result] Dave V, Brion LP, Campbell DE, Scheiner M, Raab C, Nafday SM. Splanchnic tissue oxygenation, but not brain tissue oxygenation, increases after feeds in stable preterm neonates tolerating full bolus orogastric feeding. J Perinatol. 2009 Mar;29(3):213-8. doi: 10.1038/jp.2008.189. Epub 2008 Nov 20. PMID 19020529
- [Result] Gay AN, Lazar DA, Stoll B, Naik-Mathuria B, Mushin OP, Rodriguez MA, Burrin DG, Olutoye OO. Near-infrared spectroscopy measurement of abdominal tissue oxygenation is a useful indicator of intestinal blood flow and necrotizing enterocolitis in premature piglets. J Pediatr Surg. 2011 Jun;46(6):1034-40. doi: 10.1016/j.jpedsurg.2011.03.025. PMID 21683194
- [Result] Cortez J, Gupta M, Amaram A, Pizzino J, Sawhney M, Sood BG. Noninvasive evaluation of splanchnic tissue oxygenation using near-infrared spectroscopy in preterm neonates. J Matern Fetal Neonatal Med. 2011 Apr;24(4):574-82. doi: 10.3109/14767058.2010.511335. Epub 2010 Sep 9. PMID 20828232
- [Result] Dani C, Pratesi S, Barp J, Bertini G, Gozzini E, Mele L, Parrini L. Near-infrared spectroscopy measurements of splanchnic tissue oxygenation during continuous versus intermittent feeding method in preterm infants. J Pediatr Gastroenterol Nutr. 2013 Jun;56(6):652-6. doi: 10.1097/MPG.0b013e318287e9d7. PMID 23343937